CLINICAL TRIAL: NCT06442891
Title: A Pilot Study of Self-Administered Acupressure for Fatigue Among Adolescent and Young Adult (AYA) Cancer Survivors
Brief Title: Self-Administered Relaxing Acupressure to Reduce Fatigue in Adolescent and Young Adult Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UMCC 2024.016; NCI-2024-03772 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HUM00248915 (Other: University of Michigan Comprehensive Cancer Center)
Record Dates: First submitted 2024-05-30; First posted 2024-06-04 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Acupressure; Interviews as Topic

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients are blinded to intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARM I (relaxing acupressure) (Experimental): Patients receive access to acupressure mobile application and an AcuWand on study and self-administer relaxing acupressure to 9 acupoints over 27 minutes QD for 6 weeks.
  Interventions: Procedure: Acupressure Therapy; Other: Internet-Based Intervention; Other: Interview; Other: Medical Device Usage and Evaluation; Other: Questionnaire Administration
- ARM II (sham acupressure) (Placebo Comparator): Patients receive access to acupressure mobile application and an AcuWand and self-administer sham acupressure to non-acupressure point locations over 27 minutes QD for 6 weeks.
  Interventions: Procedure: Acupressure Therapy; Other: Internet-Based Intervention; Other: Interview; Other: Medical Device Usage and Evaluation; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Acupressure Therapy — Self-administer relaxing acupressure
  Other Names: Acupressure; Ischemic Compression
  Arms: ARM I (relaxing acupressure)
Procedure: Acupressure Therapy — Self-administer sham acupressure
  Other Names: Acupressure; Ischemic Compression
  Arms: ARM II (sham acupressure)
Other: Internet-Based Intervention — Receive access to acupressure mobile app
Other: Interview — Ancillary studies
Other: Medical Device Usage and Evaluation — Receive an AcuWand
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial tests the feasibility of self-administered relaxing acupressure on fatigue in adolescent and young adult (AYA) cancer survivors. Acupressure, a type of complementary or alternative medicine, is the application of pressure or localized massage to specific sites on the body to control symptoms. Relaxing acupressure has been shown to improve cancer-related fatigue (CRF) in adults, however, less is known about the impact of relaxing acupressure on CRF in AYA cancer survivors."

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the feasibility of implementing a randomized controlled trial of a six-week, self-administered relaxing acupressure intervention in AYA cancer survivors with clinically relevant CRF.

SECONDARY OBJECTIVE:

I. Explore participants' perspectives of acceptability and satisfaction with the six-week acupressure interventions using semi-structured interviews.

EXPLORATORY OBJECTIVE:

I. Determine the preliminary efficacy of a six-week, virtual, self-administered relaxing acupressure intervention on clinically significant changes in CRF in post-treatment AYA cancer survivors.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive access to an acupressure mobile application and an AcuWand on study and self-administer relaxing acupressure to 9 acupoints over 27 minutes once daily (QD) for 6 weeks.

ARM II: Patients receive access to an acupressure mobile application and an AcuWand and self-administer sham acupressure to non-acupressure point locations over 27 minutes QD for 6 weeks.

Enrollment was increased to 45.

ELIGIBILITY:
Inclusion Criteria:

* 15 - 39 years old
* At least three months post cancer treatment (e.g., surgery, radiation or chemotherapy). Participants receiving maintenance hormonal or targeted therapies will be allowed to enroll as determined by the study investigator
* Report clinically relevant fatigue in the past seven days (Patient Reported Outcomes Measurement Information Systems [PROMIS] Fatigue 4a scores ≥ 55)
* Speak / read English
* CRF started at or after the diagnosis of cancer
* Completed cancer treatment within the past five years

Exclusion Criteria:

* Diagnosis of untreated anemia, mood disorder, or hypothyroidism
* Plan to begin new pharmacological, psychological, or other treatments (i.e., physical therapy or dietary supplements) for CRF during the study. Although, participants may continue usual treatments for CRF if the treatments were initiated at least eight weeks prior to study enrollment, and the dose has not changed
* Plan to become pregnant or lactating during the study period
* Received acupressure or acupuncture in the past year

Ages: 15 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-22 (Actual); Study Completion 2025-12-22 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | Up to 2 years
  Self-administered acupressure implementation will be feasible if all participants are recruited over 2 years. Descriptive statistics will be used to summarize recruitment rate.
Adherence | At 6 weeks
  Self-administered acupressure implementation will be feasible if 60% of participants complete the baseline and 6-week patient-reported measures and if 60% of acupressure group participants self-report acupressure practice for at least 27 minutes on at least 3 days per week. Descriptive statistics will be used to summarize adherence.
Satisfaction | Up to week 10
  Interview data will be analyzed using inductive content analysis. Perspectives of the intervention will be analyzed using inductive content analysis.
Change in fatigue | At baseline and up to week 10
  Measured using the Patient Reported Outcomes Measurement Information Systems Fatigue 4a questionnaire. Results are continuously scaled and appropriately analyzed by Gaussian-based statistical models. Change in fatigue will be analyzed using a Full Information Maximum Likelihood mixed-effects linear regression model. Specifically, change from baseline will be evaluated by including fixed-effects coefficients for time, treatment, and the important interaction effects that will determine whether changes from baseline are greater in the relaxing acupressure group, relative to controls. Random Y-intercepts in the model will be incorporated to accommodate the nesting of repeated observations within subject. Change in fatigue will be analyzed using a Full Information Maximum Likelihood mixed-effects linear regression model.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Knoerl, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided